CLINICAL TRIAL: NCT04770051
Title: Percutaneous Inferior Cervical Sympathetic Block for Treatment of Refractory Ventricular Tachycardia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of resources to conduct study.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Adnan Qureshi, Professor of Neurology, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020904
Record Dates: First submitted 2021-01-19; First posted 2021-02-25 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Percutaneous inferior cervical sympathetic block (Experimental): The procedure will be performed while the patient was awake and under fluoroscopic guidance. A total of 3 ml of 1% lidocaine will be infiltrated to anesthetize the skin and subcutaneous tissues down to the left common carotid artery. A 22 gauge × 3.5 inch BD™ Quincke spinal needle will be introduced at the level of the body of the sixth cervical vertebra, medial to the left common carotid artery. The needle will be advanced until it reached the junction between the body and transverse process of the sixth cervical vertebra. Contrast injection will be used to demonstrate the position of the needle anterior to the paravertebral muscles, with spread along the axis of the interfascial compartment (Figure 1). A total of 20 ml of 0.25% bupivacaine (Marcaine, Hospira, Lake Forest, IL) will be injected over 10 min through the needle. The effectiveness of sympathetic blockade will be confirmed by postprocedure development of ptosis and miosis in the left eye.
  Interventions: Procedure: Percutaneous inferior cervical sympathetic block

INTERVENTIONS:
Procedure: Percutaneous inferior cervical sympathetic block — The procedure will be performed while the patient was awake and under fluoroscopic guidance. A total of 3 ml of 1% lidocaine will be infiltrated to anesthetize the skin and subcutaneous tissues down to the left common carotid artery. A 22 gauge × 3.5 inch BD™ Quincke spinal needle will be introduced at the level of the body of the sixth cervical vertebra, medial to the left common carotid artery. The needle will be advanced until it reached the junction between the body and transverse process of the sixth cervical vertebra. Contrast injection will be used to demonstrate the position of the needle anterior to the paravertebral muscles, with spread along the axis of the interfascial compartment (Figure 1). A total of 20 ml of 0.25% bupivacaine (Marcaine, Hospira, Lake Forest, IL) will be injected over 10 min through the needle. The effectiveness of sympathetic blockade will be confirmed by postprocedure development of ptosis and miosis in the left eye.

SUMMARY:
The purpose of this research study is to examine the effect of percutaneous inferior cervical sympathetic block on life threatening abnormal heart rhythms called ventricular tachycardia or ventricular fibrillation that can lead to sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

1. Appropriate ICD shock for ventricular tachycardia (VT) after at least one catheter ablation of VT procedure, OR appropriate ICD shock for VT but not a candidate for catheter ablation of VT (i.e. patients with presence polymorphic VT or ventricular fibrillation, LV thrombus, VT arising from an inaccessible myocardial location).
2. Presence of structural heart disease as defined as EF ≤ 50%, presence of ventricular scar as detected by imaging modalities or electroanatomic mapping, hypertrophic cardiomyopathy, cardiac sarcoidosis, or arrhythmogenic right ventricular cardiomyopathy.
3. Patient is taking at least one anti-arrhythmic drug or has documented intolerance or toxicity to at least one anti-arrhythmic drug.
4. Age greater than 18 years old.
5. Able and willing to comply with all pre- and follow-up testing and requirements.
6. Provision of signed informed consent and stated willingness to comply with all study procedures for duration of the study.

Exclusion Criteria:

1. Active ongoing cardiac ischemia as assessed by: EKG, cardiac enzymes, symptoms, coronary angiography with evidence of significant epicardial coronary stenosis (>70%), or stress testing. (Note: positive troponin assay due to ICD shocks is not an exclusion criterion).
2. Any medical or non-medical condition likely to prevent completion of trial.
3. Contraindication to cardiac sympathetic denervation (i.e. single-lung ventilation, severe pulmonary disease, or severe pulmonary hypertension) or previous cardiac sympathetic denervation procedure.
4. Left ventricular assist device or status post orthotopic heart transplantation
5. Severe thrombocytopenia (platelets < 50,000) or coagulopathy (INR > 2.0) that is not due to medications or a reversible cause.
6. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal).
7. Unable or unwilling to comply with protocol requirements.
8. NYHA class IV heart failure symptoms.
9. Known channelopathy such as long QT syndrome and catecholaminergic polymorphic VT.
10. Presentation with slow VT (VT rate < 150 bpm).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Freedom from implantable cardioverter-defibrillator shock | 3 months
  Zero number of required cardioverter-defibrillator shocks in the patient's medical records

IPD SHARING:
Plan to Share IPD: No